CLINICAL TRIAL: NCT02480556
Title: Comparing Blood Loss Between Manual Separation & Conservative Management for Removal of the Placenta During Caesarean Section; a Randomized Controlled Study
Brief Title: Comparing Blood Loss During Caesarean Section Between Manual Separation of Placenta & Conservative Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Lecturer of Obstetrics & gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A22062015
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2015-08

CONDITIONS: Haemorrhage
Keywords: blood loss; caesarean section ; manual placental separation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): manual seperation of the placenta
  Interventions: Procedure: manual seperation of the placenta
- Group B (Active Comparator): Conservative separation of placenta
  Interventions: Procedure: Conservative separation of placenta

INTERVENTIONS:
Procedure: manual seperation of the placenta — manual separation of the placenta will be done immediately after fetal extraction & cord clamping, where the fingers of the surgeon will be insinuated between the margin of the placenta and the uterine cavity, then by sawing movement and controlled traction by the other hand till placenta is separated from the uterine cavity
  Arms: Group A
Procedure: Conservative separation of placenta — Conservative separation of placenta:
  in group B but following fetal extraction and cord clamping, the placenta will be left insitu & uterus is massaged awaiting spontaneous placental separation
  Arms: Group B

SUMMARY:
to compare the blood loss during caesarean section between two different methods of separating the placenta after fetal extraction, keeping in mind that most blood loss occurs after placental separation.

DETAILED DESCRIPTION:
We are planning a study of a continuous response variable from independent control and experimental subjects with 1 control(s) per experimental subject. In a previous study1 the response within each subject group was normally distributed with standard deviation up to 272. If the true difference in the experimental and control means is 37, we will need to study 249 experimental subjects and 249 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.5. To allow for 15% drop, the sample on each arm will be increased to 287.

After approval of the ethical & scientific committee of the obstetrics & gynecology department, Kasr Alainy Hospital, Cairo University. A randomized controlled trial involving at least 574 patients will be undertaken in which, all patients will be randomized in to two groups, with a closed envelope system containing equal number allocations for both groups (1:1 bias) by the operating room nurse. Informed consent will be taken from all patients before caesarean section.

Group A will contain 287 patients in which manual separation of the placenta will be done immediately after fetal extraction & cord clamping, where the fingers of the surgeon will be insinuated between the margin of the placenta and the uterine cavity, then by sawing movement and controlled traction by the other hand till placenta is separated from the uterine cavity. Group B will also contain 287 patients but following fetal extraction and cord clamping, the placenta will be left insitu & uterus is massaged awaiting spontaneous placental separation.

In both groups a uterotonic agent Oxytocin 5IU( syntocinon® Sandoz Pharmaceuticals Corporation East Hanover, New Jersey) will be given I.V in 250 ml ringer solution immediately after cord clamping, and the uterus is exteriorized,& the caesarean is performed by surgeons of equal training level (Senior residants). Any serious tears or extensions into the lower uterine segment, along with any major bleeding points on the suture line will be repaired before attending to the placenta in both groups to prevent any serious blood loss before placental separation, which will cause the results to be biased & increase the risk of major hemorrhage for the patient. The blood lost will be measured by recording the fluid in the suction apparatus before and after placental separation, keeping in mind that most fluid in the apparatus before fetal extraction was amniotic fluid and therefore will be deducted from the total. The net amount of fluid in the suction apparatus will be added the volume of fluid collected from blood soaked sterilized towels used after fetal extraction and the under buttocks drapes placed under the patient.

The volume of fluid collected in soaked materials will be calculated according to (2) AWHONN Practice Brief Number 1, where the dry weight of these materials in grams before the operation is recorded and subtracted from the soaked weight & converted to milliliters. The net weight will be calculated through the following equation WET Item Gram Weight - DRY Item Gram Weight = Milliliters of Blood within the item. (2) Descriptive data was recorded along with blood loss after placental separation, and the time taken for placenta to spontaneously separate in group B. Preoperative & 6 hour postoperative hemoglobin will be recorded in both groups. All statistical calculations were done using computer program SPSS (Statistical Package for the Social Science; SPSS Inc., Chicago, IL, USA) release 15 for Microsoft Windows (2006). PS Power and Sample size calculations software, version 2.1.30 for MS windows, was used to calculate sample size (Dupont & Vanderbilt, USA)

References:

1. Gol M, Baloglu A, Aydin C, Ova L, Yensel U, Karci L.(2004): Does manual removal of the placenta affect operative blood loss during cesarean section? Eur J Obstet Gynecol Reprod Biol. 2004 Jan 15;112(1):57-60.
2. AWHONN Practice Brief (2014): Quantification of Blood Loss: AWHONN Practice Brief Number 1. JOGNN, 00, 1-3; 2014. DOI: 10.1111/1552-6909.12519.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study were healthy volunteers scheduled for Caesarean section, age range between 20-38 years

Exclusion Criteria:

* Exclusion from the study included patients with anemia, abnormal coagulation defects, multi-fetal gestation, failed progress in ongoing labour, pregnancy induced hypertension & other factors increasing risk for primary postpartum hemorrhage. Diagnosed uterine fibroid or mullerian anomalies. A maximum of 10 minutes was allowed in group B before actively removing the placenta, as a diagnosis of retained placenta and abnormal placental adhesions is probably the cause and the patient was excluded from the results

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 838 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Blood Loss | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kamel, M.D, Principal Investigator — Lecturer of obstetrics & gynecology
Locations (1):
- 11562, Ḩadā’iq al Qubbah, Cairo Governorate, Egypt

REFERENCES:
- [Background] Gol M, Baloglu A, Aydin C, Ova L, Yensel U, Karci L. Does manual removal of the placenta affect operative blood loss during cesarean section? Eur J Obstet Gynecol Reprod Biol. 2004 Jan 15;112(1):57-60. doi: 10.1016/s0301-2115(03)00278-1. PMID 14687740
- [Background] AWHONN Practice Brief (2014): Quantification of Blood Loss: AWHONN Practice Brief Number 1. JOGNN, 00, 1-3; 2014. DOI: 10.1111/1552-6909.12519.